CLINICAL TRIAL: NCT06000969
Title: Conventional Versus Ultrasound-guided Lung Recruitment Manoeuvre in Morbidly Obese Patients Underdoing Laparoscopic Bariatric Surgery: Prospective Randomized Clinical Study
Brief Title: Lung Recruitment Manoeuvre in Morbidly Obese Patients Underdoing Laparoscopic Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sameh Abdelkhalik Ahmed Ismaiel, Assistant Professor of Anesthesia and Intensive Care, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 36264MD12
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Bariatric Surgery; Obesity, Morbid
Keywords: Morbidly obese, Bariatric surgery, Lung recruitment
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated in one of the two equal groups using a computer-generated table of random numbers to :-
  * Conventional group (group C); 30 patients:
  * Ultrasound-guided group (group US); 30 patients:
Who Masked: Participant, Outcomes Assessor
Masking Description: * The participants will be kept blind through the use of ultrasound assessment in both groups.
  * Outcome assessors will be blinded as they will be anesthesia resident and nurse not participating in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional group (group C) (Experimental): Patients will be shifted to 100% Oxygen then; the recruitment maneuver will be performed by manual inflation with a pressure of 30 cmH2O for 30 seconds.
  Interventions: Device: Lung Recruitment Conventional
- Ultrasound-guided group (group US) (Experimental): Patients will be shifted to 100% Oxygen then; the recruitment maneuver will be performed under the direct real-time guidance of ultrasound if atelectasis (defined as LUS of ≥ 2 for any of the 12 regions) is present. This will be done by manual inflation with a pressure of 10 cmH2O for 10 seconds, increased 10 cmH2O every 10 seconds until no collapsed areas are visible on the ultrasound, the maximum airway pressure will be limited to 40 cmH2O. This could be repeated if needed.
  Interventions: Device: Lung Recruitment Ultrasound

INTERVENTIONS:
Device: Lung Recruitment Conventional — the recruitment maneuver will be performed by manual inflation with a pressure of 30 cmH2O for 30 seconds.
  Arms: Conventional group (group C)
Device: Lung Recruitment Ultrasound — the recruitment maneuver will be performed under the direct real-time guidance of ultrasound if atelectasis (defined as LUS of ≥ 2 for any of the 12 regions) is present. This will be done by manual inflation with a pressure of 10 cmH2O for 10 seconds, increased 10 cmH2O every 10 seconds until no collapsed areas are visible on the ultrasound, the maximum airway pressure will be limited to 40 cmH2O. This could be repeated if needed.
  Arms: Ultrasound-guided group (group US)

SUMMARY:
Lung ultrasonography is an easy-to-use, portable, non-invasive, visual, and non-radiative technique that has been widely used in clinical monitoring and diagnosis.

Many studies have demonstrated that pulmonary ultrasonography can evaluate the degree of aeration loss and diagnose atelectasis accurately by using a validated semiquantitative score in the perioperative period, and lung ultrasonic imaging can be conducive to confirming the effects of lung recruitment manoeuvres.

This clinical trial suggested that the use of ultrasound-guided recruitment maneuver in morbidly obese patients scheduled for laparoscopic bariatric surgery can improve the lung aeration, decrease the incidence of basal lung atelectasis, decrease the incidence of intraoperative& postoperative oxygen desaturation, and reduce the incidence of post operative pulmonary complications.

The aim of this prospective randomized clinical study is to compare the conventional recruitment manoeuvre and ultrasound-guided recruitment manoeuvre in morbidly obese patients scheduled for laparoscopic bariatric surgery.

DETAILED DESCRIPTION:
* This prospective randomized clinical double-blinded study will be carried out at Anesthesiology Department in Tanta University Hospitals for one year from August 2023 to August 2024 after approval from our institutional ethical committee. All enrolled patients will sign an informed written consent to participate in the study.
* Every patient will receive an explanation of the purpose of the study and have secret code number to ensure privacy and confidentiality, all given data will be used for scientific purposes only.
* Any unexpected risks encountered during the research will be cleared to the participants, as well as to the Ethical Committee on time. The risk at the study includes increased risk of bradycardia and hypotension that will be managed by adequate monitoring, atropine, IV fluids, and ephedrine.

-Patients will be randomly allocated in one of the two equal groups using a computer-generated table of random numbers to :-

• Conventional group (group C); 30 patients: Patients will be shifted to 100% Oxygen then; the recruitment maneuver will be performed by manual inflation with a pressure of 30 cmH2O for 30 seconds.

• Ultrasound-guided group (group US); 30 patients: Patients will be shifted to 100% Oxygen then; the recruitment maneuver will be performed under the direct real-time guidance of ultrasound if atelectasis (defined as LUS of ≥ 2 for any of the 12 regions) is present. This will be done by manual inflation with a pressure of 10 cmH2O for 10 seconds, increased 10 cmH2O every 10 seconds until no collapsed areas are visible on the ultrasound, the maximum airway pressure will be limited to 40 cmH2O. This could be repeated if needed.

-Anesthesia technique

I-Preoperative assessment:

▪ All patients will be assessed preoperatively at the Anesthesia Clinic through history, physical examination and requesting the appropriate investigations.

II-In the Holding Area:

* Patient counselling regarding anesthesia technique and surgery.
* Secured IV line.

III- In the Operation Room:

* Standard Monitoring: On arrival of the patient to the operating theater and before induction of anesthesia, all standard monitors will be applied, including heart rate (HR), ECG, oxygen saturation (SpO2), end-tidal CO2, non-invasive blood pressure, and temperature.
* Induction of anesthesia: all patients will be pre-oxygenated with 80% oxygen for 3 minutes before induction. Anesthesia will be induced by slowly titrating doses of intravenous fentanyl (2 ug/kg of lean body weight) and propofol (1 mg/kg of lean body weight). Intubation will be facilitated with atracurium (0.5 mg/kg of lean body weight). Anesthesia will be maintained with atracurium, isoflurane of 1 MAC and fraction inspired Oxygen of 0.5 for each patient.
* Mechanical ventilation protocol: patients will receive the standard ventilation protocol as follows: volume-controlled ventilation mode, with a tidal volume of 4-6 mL/kg of predicted body weight, inspiratory: expiratory ratio 1: 2, PEEP 5 cmH2O, initial respiratory rate is 12/m then adjusted to keep end-tidal carbon dioxide tension (EtCO2) between 35- and 40-mm Hg, and inspired oxygen fraction of 0.5 with total gas flow 1L/m. The patients and investigators who will be responsible for assessing the primary outcomes will be blinded to study group assignment. However, the attending anesthesiologists, intraoperative nursing staff, and intraoperative assessors will not be blinded to study group assignment.
* Positioning and pneumoperitoneum: the patients will be put in reverse trendelenburg position, 30°C head-up position slowly, the position will be kept until the end of surgery.

Intraabdominal pressure will be maintained between 12 ± 3 cmH2O during surgery.

▪ Lung ultrasound examination: will be done: After the induction of anaesthesia (time point T1). After pneumoperitoneum (time point T2). At the end of surgery (before administrating reversal agents for neuromuscular blockade; (time point T3).

* Lung recruitment: recruitment maneuver will be performed in each group as described before after every intraoperative lung ultrasound examination. Intra-abdominal pressure will be recorded. If hypotension (MAP<65mmhg), bradycardia (heart rate<50/m.) or oxygen desaturation (spO2<95%) has been occurred, rescue strategy will be applied as described later.
* Rescue strategy for oxygen desaturation: In both groups, when SpO2 decreased to 95% or lower, the following rescue ventilation strategies will be performed in a stepwise manner (i.e., if SpO2 did not increase after a step, then the following step was applied; otherwise, no further steps were applied).

Steps were performed according to the following order:

* Step (1), three rounds of recruitment maneuvers with a pressure of 30 cmH2O for 10 s.
* Step (2), three rounds of recruitment maneuvers with a pressure of 35 cmH2O for 10 s.
* Step (3), increase FIO2 to 1.0. If SpO2 did not increase after all three rescue strategies, the ventilation strategies could be modified according to the attending anesthesiologist's judgement.

ELIGIBILITY:
Inclusion Criteria:

* adult morbidly obese patients of BMI more than 40, scheduled for laparoscopic bariatric surgery

Exclusion Criteria:

* Patient refusal
* Patients with history of severe obstructive or restrictive pulmonary disease.
* Patients with severe obstructive sleep apnea (OSA).
* Presence of emphysematous lung bullae.
* Decompensated cardiac disease (NYHA class 3 or 4).
* Patients with uncontrolled hepatic or renal disorders.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2023-08-14 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
the change of Lung Ultrasound Score | 2 hours
  Assessment of the changes in the lung ultrasound score

SECONDARY OUTCOMES:
The incidence of atelectasis | 2 hours
  defined as LUS of ≥ 2 for any of the 12 regions
The incidence of intra-operative desaturation | 3 hours
  defined as an SpO2 <95%

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Ismaiel, M.D, Principal Investigator — Assistant Professor of Anesthesia and Intensive Care, Tanta University
Locations (2):
- Egypt (2):
  - Tanta University, Tanta, Algharbia
  - Tanta University hospitals, Tanta

IPD SHARING:
Plan to Share IPD: Yes
The IPD will be available with the principle investigator within 6 months after publishing the study.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: within 6 months after publishing the study.
Access Criteria: Contact samehabdelkhalik1982@gmail.com